CLINICAL TRIAL: NCT01635088
Title: Onset and Duration of Action of Mometasone Inhalation Powder as Measured by Oscillometry Versus Spirometry
Brief Title: Onset and Duration of Mometasone by Oscillometry and Spirometry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Allergy and Asthma Medical Group, Inc. (Other)
Responsible Party: Principal Investigator, Sheldon Spector, MD, President, California Allergy and Asthma Medical Group, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05285
Record Dates: First submitted 2012-06-29; First posted 2012-07-06 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: Asthma; FEV1 and IOS change after mometasone for asthma
MeSH Terms: conditions — Asthma | interventions — Oscillometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate 220 vs. Mometasone furoate 440 (Other)
  Interventions: Drug: Mometasone furoate 220; Drug: Mometasone furoate 440
- Mometasone 220 mcg vs. 440 mcg (Active Comparator): Inhaled steroid
  Interventions: Device: KoKo Spirometry; Device: Oscillometry

INTERVENTIONS:
Drug: Mometasone furoate 220 — dry powder inhaler QD for 28-43 days
  Arms: Mometasone furoate 220 vs. Mometasone furoate 440
Device: KoKo Spirometry
  Other Names: by Nspire
  Arms: Mometasone 220 mcg vs. 440 mcg
Drug: Mometasone furoate 440 — dry powder inhaler QD for 28-43 days
  Arms: Mometasone furoate 220 vs. Mometasone furoate 440
Device: Oscillometry
  Other Names: by Jaeger, MS IOS Digital
  Arms: Mometasone 220 mcg vs. 440 mcg

SUMMARY:
Inhaled corticosteroids (ICS) are appreciated for their long term anti-inflammatory effects in chronic asthma. However, they also have largely unappreciated early effects when initiated as a controller therapy in a steroid-naïve population. Impulse oscillometry might reveal such an early effect better than spirometry. The investigators sought to examine the onset of action and sustained effects over 4 weeks treatment of mometasone furoate as measured by Impulse Oscillometry System (IOS) versus spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years inclusive.
* Written informed consent (conducted according to the GCP and ICH guidelines) to participate in the study. Ability to comply with all study requirements.
* Mild to moderate persistent asthma with symptoms at least 2 times per week, managed by as-needed SABA only.
* A 35% or greater improvement in small airway dysfunction defined by IOS AX after inhaled SABA.
* Allergic response to one or more common allergens at screening via skin test.
* Male, or female of childbearing potential using a medically approved birth control method.
* Evidence of SAD manifested by an index of peripheral airway reactance of > 10.5 cm H2O/L (3 times the upper limit of adult normal).
* Symptoms of airflow obstruction (i.e. dyspnea on exertion greater than peers at similar exercise levels, wheeze, or cough > 3 weeks without respiratory infection, or nocturnal dyspnea, and use of SABA > 2 times per week)

Exclusion Criteria:

* Subjects with severe persistent asthma and/or subjects taking inhaled or systemic corticosteroids or long acting beta agonists (LABA).
* Subjects < 18 years of age or > 65 years.
* Pregnant or lactating females.
* History of diabetes.
* Acute infections within 4 weeks prior to Screening.
* Concurrent medical condition that might interfere with the interpretation of efficacy and safety data during the study.
* Contraindications and warnings according to the specific label for Asmanex.
* Chronic inhaled or systemic corticosteroid treatment (> 7 consecutive days of treatment) within 30 days prior to Screening.
* Investigational drug treatment within 30 days prior to Screening. Treatment with any drug with a known and frequent toxicity to a major organ system within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
IOS | 4 weeks
  Measurement of pulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon L Spector, MD, Principal Investigator — California Allergy and Asthma Medical Group, Inc.
Locations (1):
- California Allergy and Asthma Medical Group, Inc., Los Angeles, California, United States